CLINICAL TRIAL: NCT03370653
Title: A Phase IIa Study to Investigate Safety, Pharmacokinetics, and Efficacy of Odiparcil in Patients 16 Years and Above With Mucopolysaccharidosis (MPS) Type VI
Brief Title: A Study in MPS VI to Assess Safety and Efficacy of Odiparcil
Acronym: iMProveS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVA_01_ODI_HMPS_17_002
Record Dates: First submitted 2017-11-23; First posted 2017-12-12 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Mucopolysaccharidosis VI
Keywords: MPS VI; Lysosomal disease; Glycoaminoglycans (GAG); Odiparcil
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — odiparcil

STUDY DESIGN:
Intervention Model Description: Preliminary safety assessment (N=2): an open-label, escalating dose (2 doses) study.
  Core study: conducted on 2 populations in parallel:
  * A first cohort (N=18): MPS VI patients receiving ERT assigned in 3 arms:
    * Placebo (N=6)
    * Odiparcil 500 mg per day (250 mg BID) (N=6)
    * Odiparcil 1000 mg per day (500 mg BID) (N=6).
  * A second cohort (N=6): MPS VI patients not receiving ERT (odiparcil 1000 mg per day (500 mg BID)).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Double-blind - odiparcil 1000 mg per day (Experimental): 2 tablets of odiparcil 250 mg per os, twice daily (BID)
  Interventions: Drug: Odiparcil
- Double-blind - odiparcil 500 mg per day (Experimental): 1 tablet of placebo and 1 tablet of odiparcil 250 mg per os, twice daily (BID)
  Interventions: Drug: Odiparcil; Other: Placebo
- Double-blind - placebo (Placebo Comparator): 2 tablets of placebo per os, twice daily (BID)
  Interventions: Other: Placebo
- Open Label - odiparcil 1000 mg per day (Experimental): 2 tablets of odiparcil 250 mg per os, twice daily (BID)
  Interventions: Drug: Odiparcil

INTERVENTIONS:
Drug: Odiparcil — Investigational product: odiparcil 250 mg tablets
  Arms: Double-blind - odiparcil 1000 mg per day; Double-blind - odiparcil 500 mg per day; Open Label - odiparcil 1000 mg per day
Other: Placebo — Comparator: placebo tablets similar to odiparcil 250 mg tablets
  Arms: Double-blind - odiparcil 500 mg per day; Double-blind - placebo

SUMMARY:
Mucopolysaccharidoses (MPS) are a group of rare inherited disorders characterized by a deficiency of lysosomal enzymes responsible for the normal degradation of glycosaminoglycans (GAGs). Medical need for treatment of MPS is still very high due to the poor penetration of the recombinant enzymes into the blood brain barrier as well as the ocular barriers and into tissues that are poorly vascularized, such as cartilages and bones. Odiparcil is an orally active compound that allows the synthesis of soluble glycosaminoglycans (GAGs), mainly chondroitin sulfate (CS) and dermatane sulfate (DS). The neosynthesized solubles GAGs are then excreted in urine. By diverting endogenous GAG synthesis to the synthesis of soluble odiparcil linked GAGs, odiparcil should decrease the intracellular pool of GAGs and consequently decrease the lysosomal GAG accumulation.

The primary objective of the study is to assess the safety and efficacy of two doses of odiparcil in MPS VI patients and to provide evidence to enable the selection of the relevant dose of odiparcil for phase III study. The secondary objective of this study is to characterize the dose response, PK and PD of odiparcil.

DETAILED DESCRIPTION:
Study design: This phase IIa study consists of 2 parts performed sequentially: a preliminary safety assessment followed by the core study with a double-blind, randomized, dose-ranged cohort of patients receiving Enzyme Replacement Therapy (ERT) and an open-label cohort of patients not receiving ERT.

Preliminary safety assessment (N=2): open-label, escalating dose (2 doses) study. If acceptable safety profile is achieved, patients will be then included in the open-label arm of the core study.

Core study

Core study will be conducted on 2 populations in parallel:

* A first cohort (N=18): MPS VI patients receiving ERT assigned in 3 arms:

  * Placebo (N=6)
  * Odiparcil 500 mg per day (250 mg BID) (N=6)
  * Odiparcil 1000 mg per day (500 mg BID) (N=6).
* A second cohort (N=6): MPS VI patient not receiving ERT (odiparcil 1000 mg per day (500 mg BID)).

Study duration: The overall study duration will be 20 months, including the 10-month enrolment period.

For each patient, the study duration will be:

* Preliminary safety assessment: 6 weeks including a 4-week run-in period followed by 2-week treatment period. Then, patients will go on treatment period in core study.
* Core study: 34 weeks including a 4-week run-in period followed by 26-week treatment period and 4-week of follow-up.

ELIGIBILITY:
1. Male or female gender.
2. Age ≥16 years.
3. Diagnosis of MPS VI, demonstrated by a reduced Arylsulfatase B (ARSB) activity relative to the normal range of the laboratory performing the assay in either white blood cells or fibroblast culture or confirmation of two known disease causing mutations in the ARSB gene.
4. Urine GAG above upper limit of normal (ULN) based on historical data.
5. Willing and able to provide written, dated, signed informed consent, or in the case of subjects age < 18 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures or study assessment.
6. Able to comply with all study procedures.
7. Women with childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy) must agree to use a highly effective method of birth control during the study and at least 4 weeks after last administration. The following can be considered to be examples of highly effective methods of contraception preferably with low user dependency:

   * Combined (estrogen and progestogen containing hormonal contraception) associated with inhibition of ovulation (oral, intravaginal, or transdermal)
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable )
   * intrauterine device (IUD)1
   * intrauterine hormone-releasing system (IUS) 1
   * Bilateral tubal occlusion1
   * Vasectomised partner1
   * Sexual abstinence These methods of contraception must be supplemented with a barrier method (preferably male condom).

Women with childbearing potential are required to have a confirmed negative blood pregnancy test before starting medication administration at baseline (V0). Women with childbearing potential agree to repeat blood pregnancy tests at visits in hospital (V2, V4, V7 and V8) and to perform urine pregnancy test before each phone call visit (V3, V5 and V6).

Inclusion criteria for ERT treated group:

1. Patients with MPS Type VI receiving enzyme replacement therapy (Naglazyme) for at least 6 months on the licensed dosage or as per local guidelines.

Inclusion criteria for not ERT treated group:

Patients with MPS Type VI not receiving enzyme replacement therapy for the following reasons:

1. Patients previously treated with ERT but have discontinued for more than 3 months either due to medical decision or personal choice
2. Patients allergic to ERT therapy
3. Patients that have had a previous hematopoietic stem cell transplant (HSCT)
4. Patients not treated with ERT i.e. treatment naïve

Exclusion criteria:

Exclusion criteria for the entire cohort:

1. Use of any investigational product or investigational medical device within 30 days prior to screening. This will include product bought over the counter specifically compounds like genistein and pentosane polysulphate which may not be considered as investigational products by patients and some health care professionals.
2. Concurrent disease or condition that would interfere with study participation or pose a safety concern for example patient with: severe cardiac insufficiency as define NYHA class > II, and severe restrictive chronic respiratory insufficiency as reflected by serum [HCO3-] ≥28 mEq/L.
3. Subjects who had surgery within 3 months before study starts, or for whom surgery is planned during study period.
4. Patient with spinal cord compression requiring surgical intervention.
5. Subjects with the following liver test anomalies: any ALT, AST > 3xULN or bilirubin >1.5xULN (except if Gilbert syndrome) at screening visit.
6. Evidence of an immunosuppressive state, including known HIV infection, agammaglubilinemias, T-Cell deficiencies.
7. Subjects with history of chronic infections, including but not limited to subjects with past history of viral hepatitis C, or B, with recent history of serious or life-threatening infection or any current signs or symptoms that may indicate infection at visit V-1 of study as per investigators clinical judgement.
8. History of malignant cancer except of cervical carcinoma in situ, basal cell carcinoma, dermatological squamous cell carcinoma.
9. Subjects with significant haematologic abnormalities, such as haemoglobin <8 g/dL, or WBC<2000 /mm3 or absolute neutrophil count <1300 /mm3, or platelet <30.000 /mm3.
10. International Normalized Ratio (INR), activated partial thromboplastin time (aPTT) or thrombin time (TT) values above the laboratory reference range at screening. For patients on anti-coagulants, they should be within their target effect on INR and be stable.
11. Any history of bleeding diathesis
12. Patient with coexistence of corneal pathologies other than corneal clouding (e.g. exposure keratopathy)
13. An unwillingness on the part of male patients to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness to use highly effective form of birth control if engaging in sexual intercourse with a woman who could become pregnant from the time of the first dose of study medication until completion of follow-up procedures.
14. An unwillingness on the part of female patients to use highly effective form of birth control2 if engaging in sexual intercourse and to have a monthly pregnancy test during treatment and until completion of follow-up procedures.
15. Pregnant or lactating women.
16. Have a known hypersensitivity to any of the ingredients or excipients of the IMP including: Microcrystalline Cellulose, Povidone, Sodium starch glycolate (type A), Magnesium stearate, Opadry™ II 85F18422

Exclusion criteria for ERT treated group:

1. Previous hematopoietic stem cell transplant (HSCT)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with modified clinical signs | 26 weeks
  Changes in physical examination and vital signs
Number of patients with modified biological values | 26 weeks
  Change from baseline in laboratory safety tests (coagulation, liver enzymes and crystalluria) 12-lead-ECG and bone biomarkers.
Incidence of AEs/SAEs | 26 weeks
  Incidence of AEs/SAEs, patient withdrawals from study due to AEs/SAEs,
12-lead ECG | 26 weeks
  Change from Baseline in ECG

SECONDARY OUTCOMES:
Mobility: 6-minute walk test | 26 weeks
  Change from baseline in 6-minute walk test
Mobility: 9-hole PEG test | 26 weeks
  Change from baseline in 9-hole PEG test
Mobility: range of motion of the shoulder | 26 weeks
  Change from baseline in range of motion of the shoulder
Pain assessment | 26 weeks
  Change from Baseline in Brief Pain Inventory (BPI)
Respiratory function | 26 weeks
  Change from Baseline in FEV1
Respiratory function | 26 weeks
  Change from Baseline in FVC
Respiratory function | 26 weeks
  Change from Baseline in MVV
Cardiac and vascular function | 26 weeks
  Change from Baseline in echocardiogram
Cardiac and vascular function | 26 weeks
  Change from Baseline in carotid intima media thickness Odiparcil concentration remaining in patient plasma 12 hours following the last intake of investigational product at visits V4 and V7. An identification of odiparcil metabolites in plasma at visit V2.
Audiology assessments | 26 weeks
  Change from Baseline in pure tone audiometry
Audiology assessments | 26 weeks
  Change from Baseline in whisper voice test
Ophthalmology assessments | 26 weeks
  Change from Baseline in corneal opacification
Ophthalmology assessments | 26 weeks
  Change from Baseline in level of retinopathy
Ophthalmology assessments | 26 weeks
  Change from Baseline in optic nerve involvement,
Ophthalmology assessments | 26 weeks
  Change from Baseline in intra-ocular pressure
Ophthalmology assessments | 26 weeks
  Change from Baseline in visual acuity
Quality of life questionnaires | 26 weeks
  Change from Baseline in EQ-5D-5L questionnaires. 5 dimensions scored on a 5-point scale will be assessed: mobility, self-care, usual activities, pain/discomfort, anxiety/depression
Quality of life questionnaires | 26 weeks
  Change from Baseline in Zarit caregiver burden questionnaires. Scale in 22 items scored on a 5-point scale with 0 = never and 5 = nearly always
Quality of life questionnaires | 26 weeks
  Change from Baseline in Fatigue Severity Scale questionnaires. 9 questions scored on a 7-point scale with 1 = strongly disagree and 7= strongly agree
Pharmacokinetics: odiparcil concentration in plasma | 12 hours
  Odiparcil concentration in plasma at visit V2 (up to 12 hours post dose).
¨Pharmacodynamics: GAG concentrations | 26 weeks
  GAG concentration in leukocytes isolated from peripheral
¨Pharmacodynamics: GAG concentrations | 26 weeks
  GAG concentrations in urine
Pharmacodynamics: GAG concentrations | 26 weeks
  GAG concentrations in skin
¨Pharmacodynamics: anti-thrombin activity IIa | 26 weeks
  Change from Baseline in anti-thrombin activity IIa in plasma
¨Pharmacodynamics: Thrombin Generation Assay (TGA) | 26 weeks
  Change from Baseline in TGA in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Derralynn HUGHES, MD, Principal Investigator — Royal Free Hospital, London UK; Julia HENNERMANN, MD, Principal Investigator — Villa Metabolica, Mainz GERMANY; Nathalie GUFFON-FOUILHOUX, MD, Principal Investigator — Hôpital Femme-Mère-Enfant; Elisa LEAO-TELES, MD, Principal Investigator — Centro Hospitalar S. João, Porto, Portugal
Locations (4):
- Hôpital Femme-Mère-Enfant, Bron, France
- Villa Metabolica, Mainz, Germany
- Centro Hospitalar S. João, Porto, Portugal
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No